CLINICAL TRIAL: NCT03030027
Title: Connecting Through Caregiving: Reappraising Intergeneration Relationships for Dementia Caregivers
Brief Title: Connecting Through Caregiving: Reappraising Intergeneration Relationships
Acronym: CTC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AFC2016
Record Dates: First submitted 2017-01-08; First posted 2017-01-24 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2017-01

CONDITIONS: Dementia
Keywords: Intergeneration; Reappraisal; Caregiving
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Connecting Through Caregiving (Experimental): This arm focuses on perspective-taking reappraisal procedures.
  Interventions: Behavioral: Connecting Through Caregiving
- Basic Skills Building (Other): This arm focuses on skill building.
  Interventions: Other: Basic Skills Building

INTERVENTIONS:
Behavioral: Connecting Through Caregiving — The Connecting Through Caregiving intervention focuses on reappraisal exercises on intergeneration relationships in caregiving, involving the following: 1) enhancing self-awareness of the caregiver, 2) developing interpersonal empathy for the care-recipient, 3) help-seeking in caregiving, 4) balancing self-care and caring and 5) negotiating action plans.
  Arms: Connecting Through Caregiving
Other: Basic Skills Building — Skill building involves: 1) monitoring activities, 2) pleasant event scheduling, 3) communicating with the care recipient, 4) communicating with family members and 5) review implementation
  Arms: Basic Skills Building

SUMMARY:
The purpose of the present study is to examine the effects of perspective-taking reappraisals on the well-being of adult-child dementia caregivers.

DETAILED DESCRIPTION:
Dementia caregiving presents a particular challenge wherein the adult child is parenting his or her parents. Facilitating relational insights, the key components of the Connecting Through Caregiving (CTC) intervention involves the following: 1) enhancing self-awareness of the caregiver, 2) developing interpersonal empathy of the care-recipient, 3) help-seeking, 4) balancing self-care and caring for others and 5) negotiating action plans. The CTC intervention is be evaluated against a basic skill training intervention consisting of scheduling pleasant events, communicating with the care recipient and other family members. Dementia caregivers providing at least 14 hours of care per week to a parent living with dementia are recruited and randomized into one the two conditions. The intervention lasts for six weeks for both conditions. Intervention in the first week consists of a home visit and a telephone follow-up. From the second to fifth week, there are weekly four telephone phone sessions. In the sixth week, there were two more telephone calls to consolidate the intervention and to review implementation plans.

ELIGIBILITY:
Inclusion Criteria:

* The study participants will be primary caregivers aged 18 or older and who have been caring for persons (aged 60 or above) with a physician diagnosis of Alzheimer's disease in the mild to moderate range as determined by the Clinical Dementia Rating Scale.
* Primary caregivers are those who have been providing unpaid care for more than 14 hours a week for at least the past three months.
* The care should involve day-to-day decision-making as well as any of the following: feeding, dressing, bathing, toileting, housework, preparing meals, medication and handling finances.
* They can be daughter/son or daughter-/son-in-law of the care recipients.

Exclusion Criteria:

* Exclusion criteria are as follows: signs of severe intellectual deficits, demonstrated suicidal ideation, exhibited evidence of psychotic disorders, hearing/ visual impairment or inability to read or speak Chinese/Cantonese fluently and severe.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-01-09 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Life Satisfaction (LS): scale | Change from Baseline LS through study completion, an average of 2 months
  Each response was rated from to 7 on each of the 5 items of the scale with higher score indicating higher level of life satisfaction
Change in Center for Epidemiologic Studies Depressive Scale (CESD) | Change from Baseline CESD through study completion, an average of 2 months
  Each response was rated from 0 to 3 on a scale of the frequency of the occurrence of the symptom in the past week. Higher scores would suggest a higher

SECONDARY OUTCOMES:
Change in Zarit Burden Interview (ZBI) | Change from Baseline ZBI through study completion, an average of 2 months
  Each of the 22 items required the caregiver to rate on a 5-point scale ranging from 0 (never) to 4 (nearly always).

CONTACTS AND LOCATIONS:
Overall Officials: Alma Au, {PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Institute of Active Ageing, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No